CLINICAL TRIAL: NCT01221506
Title: Assessment of Tumor Perfusion Changes in Response to Pazopanib in Renal Cell Carcinoma
Brief Title: Pazopanib/DCE-MRIs in Renal Cell Carcinoma (RCC)
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 34809
Record Dates: First submitted 2010-10-13; First posted 2010-10-15 (Estimated); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Carcinoma, Renal Cell
Keywords: unresectable; metastatic; clear cell renal carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell; Neoplasm Metastasis | interventions — pazopanib; Dynamic Contrast Enhanced Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Pazopanib — 800 mg PO QD x 28 days
Device: DCE-MRI and Quantitative Doppler Ultrasound — Contrast-enhanced MRI

SUMMARY:
All patients who participate in this study will receive pazopanib. Pazopanib is an oral drug (pill) that has been approved by the U.S. Food and Drug Administration (FDA) for the treatment of advanced kidney cancer. In this study, the investigators plan to learn more about the way this drug works by using special scans (MRIs and Ultrasounds) to help evaluate how this drug is working on this disease. Approximately 20 people with advanced kidney cancer will be enrolled on this study.

DETAILED DESCRIPTION:
Overall objectives PRIMARY: - Assessment of early changes in DCE-MRI and ultrasound measures of tumor perfusion in the setting of pazopanib therapy for patients with metastatic clear cell renal cell carcinoma SECONDARY: - Correlation of baseline DCE-MRI and ultrasound parameters and clinical outcome - Correlation of early (48 +/- 24 hr after treatment) changes in DCE-MRI and ultrasound parameters and clinical outcome - Correlation of baseline (and changes) in DCE-MRI and ultrasound parameters with VHL status in tumors and histocytometric analysis of endothelial cell activation in archival nephrectomy specimens - Provide an insight in the respective predictive values of DCE-MRI and US for pazopanib treatment

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Diagnosis of unresectable and/or metastatic clear cell renal cell carcinoma. 10 patients will be enrolled who have had no prior anti-angiogenic therapy; 10 patients will be enrolled who have had one prior anti-angiogenic therapy
* Prior radiation therapy to a symptomatic site of metastatic disease is allowed but patients must have discontinued/completed radiation therapy at least 2 weeks prior to entering the study, and have recovered from adverse events due to that treatment.
* ECOG performance status of 0, 1 or 2.
* Patients must have measureable disease by RECIST 1.1
* Archived tumor blocks must be provided for all subjects for correlative analysis before or during treatment with pazopanib
* Patient must have normal baseline laboratory values
* Patients must not receive any other investigational agents while onstudy.
* Patients must not be taking cytochrome P450 enzyme -inducing antiepileptic drugs (phenytoin, carbamazepine or phenobarbital), rifampin or St.Johns wort.
* Females of childbearing potential are eligible to enter and participate in this study if they have a negative pregnancy test and agree to use medically accepted contraception throughout the study

Exclusion Criteria:

* Female subjects who are pregnant or brestfeeding - Patients with active prior malignancy. Note: Subjects who have had another malignancy and have been disease-free for 3 years, or subjects with a history of completely resected non-melanomatous skin carcinoma or successfully treated in situ carcinoma are eligible.
* Patients with a history or clinical evidence of central nervous system (CNS) metastases or leptomeningeal carcinomatosis, except for individuals who have previously-treated CNS metastases, are asymptomatic, and have had no requirement for steroids or anti-seizure medication for 6 months prior to first dose of study drug. Screening with CNS imaging studies (computed tomography [CT] or magnetic resonance imaging [MRI]) is required only if clinically indicated or if the subject has a history of CNS metastases.
* Patients with clinically significant gastrointestinal abnormalities that may increase the risk for gastrointestinal bleeding
* Patients with clinically significant gastrointestinal abnormalities that may affect absorption of investigational product
* Patients the presence of uncontrolled infection.
* Patient with corrected QT interval (QTc) greater than 480 msecs using Bazetts formula
* Patients with a history of any one or more of the following cardiovascular conditions within the past 6 months: Cardiac angioplasty or stenting; Myocardial infarction; Unstable angina; Coronary artery bypass graft surgery; Symptomatic peripheral vascular disease; Class III or IV congestive heart failure, as defined by the New York Heart Association (NYHA) [See Section YYY Appendix Y for description
* Patient with poorly controlled hypertension [defined as systolic blood pressure (SBP) of greater or equal to 140 mmHg or diastolic blood pressure (DBP) of greater or equal to 90mmHg].
* Patients with a history of cerebrovascular accident including transient ischemic attack (TIA),pulmonary embolism or untreated deep venous thrombosis (DVT) within the past 6 months. Note: Subjects with recent DVT who have been treated with therapeutic anti-coagulating agents for at least 6 weeks are eligible
* Patients who have had prior major surgery or trauma within 28 days prior to first dose of study drug and/or presence of any non-healing wound, fracture, or ulcer (procedures such as catheter placement not considered to be major).
* Patients who have evidence of active bleeding or bleeding diathesis.
* Patients with known endobronchial lesions and/or lesions infiltrating major pulmonary vessels
* Patients with hemoptysis within 6 weeks of first dose of study drug.
* Patients with any serious and/or unstable pre-existing medical, psychiatric, or other condition that could interfere with subjects safety, provision of informed consent, or compliance to study procedures.
* Patients who are unable or unwilling to discontinue use of prohibited medications list in Section4.3 for at least 14 days or five half-lives of a drug (whichever is longer) prior to the first dose of study drug and for the duration of the study.
* Treatment with any of the following anti-cancer therapies: radiation therapy, surgery or tumor embolization within 14 days prior to the first dose of pazopanib; OR chemotherapy,immunotherapy, biologic therapy, investigational therapy or hormonal therapy within 14 days prior to the first dose of pazopanib. Treatment with prior sorafenib, sunitinib, temsirolimus or everolimus is allowed but must be discontinued at least 5 days prior to beginning pazopanib.
* Patient who have any ongoing toxicity from prior anti-cancer therapy that is greater than Grade 1 and/or that is progressing in severity, except alopecia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-10 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Evaluate Early Changes in DCE-MRI | 12 weeks
  To evaluate early changes in DCE-MRI measures of tumor vascular permeability after treatment with pazopanib.

SECONDARY OUTCOMES:
Correlating Baseline DCE-MRI and early changes in DCE-MRI with other measures of treatment effectiveness
  Correlating baseline DCE-MRI and early changes in DCE-MRI with other measures of treatment effectiveness, including clinical outcomes and histologic measures of tumor angiogenesis.

CONTACTS AND LOCATIONS:
Overall Officials: Naomi Haas, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States